CLINICAL TRIAL: NCT03737903
Title: Preoperative Use of Wrist-worn Accelerometers to Measure Physical Activity in High-risk Elderly Patients
Brief Title: Understanding Pre-operative Activity Levels in Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Joanne Outtrim (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor-Investigator, Joanne Outtrim, Senior Research Nurse, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: A094782; 238840 (Other: IRAS Number)
Record Dates: First submitted 2018-05-08; First posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Surgery; Physical Activity; Aging
Keywords: Frail elderly; Accelerometer; Preoperative assessment
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim to determine whether a wrist-worn accelerometer device is able to objectively measure physical activity, and whether it is an acceptable process for high-risk elderly patients prior to planned surgery. Accelerometers measure physical activity in 'counts' of activity, enabling them to record the total amount of activity in a given time period (e.g. number of steps per day), and also the time spent in various levels of intensity of activity. The investigators will ask study participants to wear an accelerometer around their wrist (like a wristwatch) for up to 14 days prior to their surgery. Participants will receive the same care as non-participants. Part of this routine medical care includes a preoperative review by a multidisciplinary team including specific personalised advice to optimise physical activity before surgery. The investigators will measure the impact that this existing intervention has on physical activity levels. Being more physically active is good for our health, and may be associated with a better recovery from surgery. In the future there may be methods of improving physical activity in the period of time before patients' surgery, which may improve their recovery from surgery.

In order to study this further, the investigators first need a robust and objective way of measuring physical activity. In current practice patients are asked to estimate how physically active they are on a day-to-day basis. This relies on how well they remember, and how good they are at getting it right and may not be accurate. The wrist-worn accelerometer is an objective method of measuring physical activity in patients, which not only offers greater understanding of the physical activity levels of elderly patients before a variety of operations, but also offers the opportunity to measure the impact of existing and potential future interventions to modify physical activity in the preoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 65 years or above
* Rockwood frailty score of ≥4
* Listed for elective major or complex surgery at Cambridge University Hospitals NHS Foundation Trust
* Capacity to consent and complete activity questionnaires
* Willing and able to wear accelerometer around wrist

Exclusion Criteria:

* Does not meet the inclusion criteria
* Participant refusal
* PRIME clinic appointment scheduled less than 72hrs after the nurse led pre-assessment clinic

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The investigators are aiming to recruit approximately 50 high-risk patients aged 65 years and above, prior to major or complex elective surgery.
  "High-risk" is determined by Rockwood Clinical Frailty Score ≥4. Major or complex surgery is defined in NICE guideline (NG45).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Measuring physical activity, defined as daily average activity-related acceleration (expressed in relative gravity, milligravity) in high risk elderly patients in the preoperative period using wrist worn accelerometers. | 2 weeks
  This will be measured using a wrist worn accelerometer device to measure daily average activity-related acceleration expressed in relative gravity, milligravity.

SECONDARY OUTCOMES:
Objective measurement of baseline physical activity levels using a wrist worn triaxial accelerometer, across different surgical specialties, thereby obtaining data on the variation in physical activity, expressed in relative gravity (milligravity). | 2 weeks
  Measurement of baseline physical activity levels using a wrist worn triaxial accelerometer, across different surgical specialties, thereby obtaining data on the variation in physical activity, expressed in relative gravity (milligravity).
Measure total daily physical activity, expressed in relative gravity (milligravity), using a wrist-worn triaxial accelerometer, before and after current preoperative intervention occuring as part of routine medical care. | 2 weeks
  Measure total daily physical activity, expressed in relative gravity (milligravity), using a wrist-worn triaxial accelerometer,for one week before and one week after current preoperative intervention occurring as part of routine medical care. This will measure any change in physical activity from baseline to one week post intervention (therefore measured over a total time period of 2 weeks) as part of routine medical care
Correlation between objectively measured physical activity and patient reported physical activity | 2 weeks
  To determine any correlation between measured physical activity (expressed in relative gravity, milligravity), and patient reported physical activity (expressed using the PASE score) measured using appropriate correlation statistics
Subjective measurement of baseline physical activity levels using validated self-reported physical activity questionnaire, across different surgical specialties. | 2 weeks
  Subjective measurement of baseline physical activity levels using validated self-reported physical activity questionnaire, across different surgical specialties, thereby obtaining data on the variation in physical activity measured by the Physical Activity Scale for the Elderly (PASE) score. PASE comprises measures of self-reported occupational, household, and leisure activities during a one-week period. Scores range from 0 to 400 with a higher score indicating a higher level of physical activity
Determine participant compliance in wearing the accelerometer device | 2 weeks
  This will be measured by recording the total wear time (in hours) of the device during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Ari Ercole, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambs, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grimes L, Outtrim JG, Griffin SJ, Ercole A. Accelerometery as a measure of modifiable physical activity in high-risk elderly preoperative patients: a prospective observational pilot study. BMJ Open. 2019 Nov 3;9(11):e032346. doi: 10.1136/bmjopen-2019-032346. PMID 31685513